CLINICAL TRIAL: NCT02817477
Title: Intranasal Ketamine for Acute Traumatic Pain in the Emergency Department: A Prospective, Randomized Clinical Trial of Efficacy and Safety
Brief Title: Intranasal Ketamine for Acute Traumatic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tel Aviv Medical Center (Other)
Responsible Party: Principal Investigator, Prof. Pinchas (Pinny) Halpern MD, Chair, Emergency Department, Tel Aviv Medical Center, Tel Aviv Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0312-11-TLV
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Acute Pain
Keywords: Intranasal Ketamine, Analgesia, Trauma, Morphine, Mass Casualty
MeSH Terms: conditions — Acute Pain; Agnosia; Wounds and Injuries | interventions — Ketamine; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IN Ketamine (Experimental): A single administration of 1 mg/kg ketamine hydrochloride delivered in an intranasal route using an atomizer
  Interventions: Drug: Ketamine Hydrochloride
- IM Morphine (Active Comparator): A single administration of 0.15 mg/kg intramuscular morphine
  Interventions: Drug: Morphine
- IV Morphine (Active Comparator): A single administration of 0.1 mg/kg slow intravascular bolus of morphine.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Delivered intranasally using an atomizer
  Arms: IN Ketamine
Drug: Morphine — Delivered either as an IM injection or a slow IV bolus
  Arms: IM Morphine; IV Morphine

SUMMARY:
Introduction: Ketamine has been well studied for its efficacy as an analgesic agent. However, intranasal (IN) administration of ketamine has only recently been studied in the emergency setting.

Objective: To elucidate the efficacy and adverse effects of a sub-dissociative dose of IN Ketamine compared to IV and IM morphine.

Methods: A single-center, randomized, prospective, parallel clinical trial of efficacy and safety of IN ketamine compared to IV and IM morphine for analgesia in the emergency department (ED). A convenience sample of 90 patients aged 18-70 experiencing moderate-severe acute traumatic pain (≥80mm on 100mm Visual Analog Scale [VAS]) were randomized to receive either 1.0mg/kg IN ketamine, 0.1mg/kg IV MO or 0.15mg/kg IM MO. Pain relief and adverse effects were recorded for 1 hour post-administration.

Primary Outcomes: The primary outcome was efficacy of IN ketamine compared to IV and IM MO, measured by "time-to-onset" (defined as a ≥15mm pain decrease on VAS), as well as time to and degree of maximal pain reduction.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-70 years, with mild to moderate blunt trauma (sustained in road, workplace and home accidents) causing moderate to severe pain (≥ 80mm score on a 100mm Visual Analog Scale=VAS) were eligible for participation in the study. Inclusion criteria also included a Glasgow Coma Score (GCS) of 15, body weight of 50-110 kg, systolic blood pressure of 90-160 mmHg, heart rate <100 bpm. Patients were also required to have an American Society of Anesthesiologists (ASA) score of 1 or 2, deny head injury, and deny regular use or use of opiates.

Exclusion Criteria:

Any analgesia received within the prior 3 hours, allergic sensitivity to morphine or ketamine, a large meal ingested within the previous hour, pregnancy, deviated nasal septum or trauma to the nose, and a history of a psychiatric condition. Despite evidence that ketamine does not exacerbate intracranial hemorrhage in patients with head trauma, patients with head injury complaining of loss of consciousness, dizziness, vomiting, or nausea were excluded as well.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness of intranasal ketamine in decreasing pain intensity [patient assessed - VAS pain score] | 1 hour post administration
  Time to achieve a clinically meaningful pain reduction was defined as the first time-point at which the patient reported 15mm of pain reduction or more. Maximal pain reduction was defined as the lowest VAS score reported by the patient over the course of follow-up. Time to maximal pain reduction was defined as the time at which the patient has the lowest VAS score over the course of the hour follow-up.

SECONDARY OUTCOMES:
adverse effects [Opiate Related Symptom Distress Scale] | 1 hour post administration
  Adverse effects were recorded at the end of one hour using the 'Opiate Related Symptom Distress Scale' and included measurements of the presence, frequency, intensity and disruptiveness of 12 common opiate side-effects. Among these were nausea, vomiting, urinary retention, constipation, difficulty concentrating, dizziness, confusion, and others.
patient satisfaction [Interview] | 1 hour post administration
  patients were asked to provide subjective comments

CONTACTS AND LOCATIONS:
Overall Officials: Pinchas Halpern, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shimonovich S, Gigi R, Shapira A, Sarig-Meth T, Nadav D, Rozenek M, West D, Halpern P. Intranasal ketamine for acute traumatic pain in the Emergency Department: a prospective, randomized clinical trial of efficacy and safety. BMC Emerg Med. 2016 Nov 9;16(1):43. doi: 10.1186/s12873-016-0107-0. PMID 27829367